CLINICAL TRIAL: NCT02037659
Title: Endoscopic Ultrasound (EUS) Gastric Variceal Bleeding Database Repository
Brief Title: Dermabond Treatment for Gastric Variceal Bleeding
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Director, Endoscopic Ulatrsound, Indiana University
Other Study IDs: Dermabond
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Gastric Varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric Varices treatment: DermaBond (glue) treatment of Gastric Varices.
  Interventions: Procedure: DermaBond treatment of Gastric Varices

INTERVENTIONS:
Procedure: DermaBond treatment of Gastric Varices — Endoscopic Ultrasound (EUS) administration of DermaBond glue to control bleeding gastric varices.
  Other Names: DermaBond: (cyanoacrylate tissue adhesive).

SUMMARY:
The purpose of having a database is to collect data related to endoscopic ultrasound procedures performed by Indiana University EUS physicians; specifically, for the treatment of gastric variceal bleeding This data will be used for research purposes only to determine the clinical impact of endoscopic ultrasound treatment of gastric variceal bleeding. The physicians will also be able to better understand the patient's condition and disease process that may lead to improved standard of care and improved patient management.

DETAILED DESCRIPTION:
Clinical outcomes research is one of the strengths of the EUS group. As a group, the physicians need a tracking system for specific treatment modalities, and data to determine the impact of endoscopic ultrasound for patients with gastric variceal bleeding. Gastric variceal bleeding is a severe complication of portal hypertension with significant morbidity and mortality with limited therapeutic options. Currently, there is no database in existence for endoscopic ultrasound clinical research for specific procedures. Also, there is limited data regarding the outcome of endoscopic sclerotherapy with cyanoacrylate in the United States.

ELIGIBILITY:
Inclusion Criteria:

Anyone receiving treatment with DermaBond for treatment gastric varices.

Exclusion Criteria:

No evidence of gastric varices.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with DermaBond for gastric varices.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-12; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
To determine the clinical impact of endoscopic ultrasound treatment of gastric variceal bleeding. | 36 months
  Patients with gastric variceal bleeding will be treated with DermaBond injection via EUS (endoscopic ultrasound). A follow-up EUS will observe the treated varices and determine if retreatment with DermaBond is necessary, or if observation alone is required.

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No